CLINICAL TRIAL: NCT05153551
Title: Pediatric Early Autism Recognition System: PEARS
Acronym: PEARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Nicole Hamp, House Officer, Developmental-Behavioral Pediatrics, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00203538
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Early diagnosis
MeSH Terms: conditions — Autism Spectrum Disorder; Disease

STUDY DESIGN:
Intervention Model Description: 30 families (30 children and 30 parents/legal guardians) to be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEARS assessment (Experimental)
  Interventions: Other: Play-based assessment (RITA-T)

INTERVENTIONS:
Other: Play-based assessment (RITA-T) — The RITA-T is a play-based assessment that involves nine different activities that can be done safely with a child seated in the exam room. After scoring the RITA-T, the PEARS PCP will immediately provide feedback to the parent regarding results and next steps.
  In addition, parents will complete certain assessments/surveys during the study to evaluate the program.

SUMMARY:
The goal of the study is to assess a new autism evaluation model that would include the addition of a Level-2 autism screener, the Rapid Interactive Screening Test for Autism in Toddlers (RITA-T), to the developmental screening already done by the child's pediatrician.

The study hypotheses:

1. The PEARS intervention will show high feasibility to primary care physicians (PCPs) and patient families.
2. The PEARS intervention will lead to increased parent activation around autism diagnosis.

ELIGIBILITY:
Inclusion Criteria- Child:

* Increased risk for Autism Spectrum Disorder (ASD) defined as:

  * positive Modified Checklist for Autism in Toddlers-Revised (MCHAT) (score greater than 3);
  * OR having a sibling or parent with ASD;
  * OR history of prematurity (gestational age less or equal 34 weeks);
  * OR other provider or parent concern for ASD.
* Child age 18-36 months

Exclusion Criteria- Child:

* previous ASD diagnosis
* previous negative ASD evaluation
* known seizure disorder
* vision impairment
* hearing impairment

Inclusion Criteria- Parent

- Parent or legal guardian of the children

Exclusion Criteria- Parent

- Not a Parent or legal guardian of the child

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Proportion of PEARS PCP visits in which PCPs report overall feasibility in regard to workflow, delivery, and administration of the RITA-T | Approximately day 7 (Time 3)
  This is based on a 6 question feasibility survey (score of 24 or greater would be considered feasible).
Percentage of parents that felt that the RITA-T visit was comfortable and useful | Approximately day 35 (time 5)
  This is based on a 5 question feasibility survey (score of 20 or greater would be considered feasible).
Change on the Parent Activation Measure for Children with Developmental Disabilities (PAM-DD) | Baseline(day 1), approximately day 35 (time 5)
  Items are scored using a 4-point a Likert-type scale (1 = disagree strongly to 4 = agree strongly). Raw scores are summed and scaled from 0 to 100 using weighted scores based on Guttman scaling. Higher scores correspond to higher activation. This 13-item measure will be administered verbally to parents at baseline and 3-4 weeks post-RITA-T assessment. Changes from baseline to follow-up will be calculated for each participant.
Qualitative data from parents semi-structured interviews | Approximately day 35 (time 5)
  The study team will analyze transcripts of parent semi-structured interviews to assess general sense of empowerment and motivation, with a focus on novel insights into the experience of parents of children undergoing a Level-2 screening instrument within the medical home.

SECONDARY OUTCOMES:
The number of days between enrollment and completed RITA-T assessment | Approximately 7-14 days
The percentage of participants that experienced scheduling and/or transportation barriers | Approximately day 35 (time 5)
  This data will be collected by the research assistants or reported by parents during the follow-up semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Hamp, MD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Michigan Medicine Briarwood Center for Women, Children, and Young Adults., Ann Arbor, Michigan
  - Michigan Medicine Brighton Health Center, Brighton, Michigan
  - Michigan Medicine Northville Health Center, Northville, Michigan

IPD SHARING:
Plan to Share IPD: No